CLINICAL TRIAL: NCT01537029
Title: Effect of Weight on the Population Pharmacokinetic Analysis of Doxorubicin and Cyclophosphamide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Collaborators: University of Texas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A11-3691
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-07

CONDITIONS: Breast Cancer; Obesity
Keywords: Breast cancer; Pharmacokinetics; Obesity; Doxorubicin; Cyclophosphamide; Weight
MeSH Terms: conditions — Breast Neoplasms; Obesity; Body Weight | interventions — Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Doxorubicin and cyclophosphamide (Experimental)
  Interventions: Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Doxorubicin — Dosed by the patient's treating physician according to local standard of care.
Drug: Cyclophosphamide — dosage form: IV, Dosage, frequency, and duration: According to local standard of care

SUMMARY:
To determine the effect of weight on doxorubicin and cyclophosphamide plasma clearance in participants who are normal weight (body mass index [BMI] < 25 kg/m2, overweight or class I obese (BMI 25-34.9 kg/m2), or class II-III obese (BMI ≥ 35 kg/m2). The hypothesis is that participants who weigh more will have higher doxorubicin and cyclophosphamide clearances than participants who weigh less. Restated, the area under the drug-concentration time profile, also known as the AUC, in participants will decrease as participant weight increases.

DETAILED DESCRIPTION:
This single site study will be conducted at the UT Southwestern Simmons Cancer Center. This study is designed to measure drug concentrations in the blood of 18 female breast cancer patients who require doxorubicin (30 minute infusion) and cylcophosphamide (30 minute infusion) as part of standard medical care. Up to a total of 40 adult female participants will be consented for the study at the cancer center. Eighteen of these participants are needed to complete the study. The others will likely be screen failures. The participants will have no more than 100 ml of blood drawn via a peripheral intravenous catheter just prior to the doxorubicin infusion, and then at 0.5, 1, 1.5, 2, 3, 4, 5, 12-24, and 24-72 h after the beginning of the doxorubicin infusion. The 5 hour blood draw is optional. The intravenous catheter will be removed when the participant is discharged from the cancer center on day 1. The participant will be asked to return to the cancer center at 12-24 and 24-72 hours to have the final 2 blood draws conducted.

The participants must be treated with Doxurubicin and Cyclophosphamide in order to participate in this pharmacokinetic analysis study.

ELIGIBILITY:
Inclusion Criteria:

* Females, age 18 years of age or older, of all racial and ethnic origins that are scheduled to receive the first cycle of a single intravenous dose of doxorubicin (30 minute infusion) and cylcophosphamide (30 minute infusion) as part of standard medical care for breast cancer. English and/or Spanish speaking participants are eligible to participate.

Exclusion Criteria:

* Pregnant or nursing or unwilling to use a reliable contraception method during the study. The effects of doxorubicin and cyclophosphamide on pregnancy are unknown. In addition, the metabolic changes that accompany pregnancy may alter the concentration-time profile of doxorubicin or cyclophosphamide, so that the pregnancy and post-partum state would be a confounding variable.
* Participants unwilling to comply with study procedures.
* CrCl < 10 ml/min
* Participants requiring peritoneal or hemodialysis
* Serum bilirubin > 1.19 mg/dL
* Receipt of the following drugs that: a) Alter doxorubicin concentrations: carbamazepine, cyclosporine, fosphenytoin, paclitaxel, phenytoin, sorafenib, valspodar, verapamil; b) Alter cyclophosphamide concentrations: cyclosporine, nevirapine, ondansetron; c) All other drugs will be reviewed during screening of the patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Hall, PharmD, Principal Investigator — Texas Tech University HSC
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hall RG 2nd, Liu S, Pai MP, Putnam WC, Subramaniyan I, Kallem R, Haley B. Impact of obesity on doxorubicin pharmacokinetics in women with breast cancer. J Oncol Pharm Pract. 2025 Mar 13:10781552251326045. doi: 10.1177/10781552251326045. Online ahead of print. PMID 40080880

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Doxorubicin and Cyclophosphamide
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Doxorubicin and Cyclophosphamide
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Clearance (Cl) for Doxorubicin and Cyclophosphamide
Description: Cyclophosphamide analysis was not possible due to rapid drug degradation
Time Frame: 0-48 hours
Measure: Median (Full Range); unit: L/hr
Arm/Group | Doxorubicin and Cyclophosphamide
Number analyzed (Participants) | 13
L/hr | 1.85 [0.84 to 4.23]

ADVERSE EVENTS:
Time Frame: Pre-dose until last blood draw (24 to 48 hours was the last time point if participant completed all blood draws)
Arm/Group | Doxorubicin and Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No